CLINICAL TRIAL: NCT06018103
Title: MBCT-vision to Treat Visual Snow Syndrome: a Randomized Controlled Trial
Brief Title: MBCT-vision VSS RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 328749
Record Dates: First submitted 2023-08-25; First posted 2023-08-30 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Visual Snow Syndrome
Keywords: Visual Snow Syndrome; Mindfulness
MeSH Terms: conditions — visual snow syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial of two groups: Treatment (MBCT-vision), or Control (wait-list, standard of care)
Who Masked: Outcomes Assessor
Masking Description: Statistician performing the analysis will be masked. It is not possible to mask the participant nor the investigator due to the nature of the intervention (group learning programme on mindfulness)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): 8-week online group learning course of the MBCT-vision programme
  Interventions: Behavioral: MBCT-vision
- Control (No Intervention): wait-list control (standard care, no research intervention)

INTERVENTIONS:
Behavioral: MBCT-vision — 8-week mindfulness group learning course, using Mindfulness Based Cognitive Therapy customised for visual symptoms (MBCT-vision). Participants meet once weekly only, with daily home practice between sessions.
  Arms: Treatment

SUMMARY:
Visual Snow Syndrome (VSS) is a neurological condition with bran network dysregulation involving the visual pathway. This is a research trial comparing the effect of an 8-week mindfulness-based intervention via a group-learning course, the MBCT-vision programme, to treat Visual Snow Syndrome, compared to people on a standard care (wait-list control). Participants will be randomly allocated to either the Treatment group (MBCT-vision), or the Control group (wait-list control). After a waiting period, people allocated to the Control group will also be offered the MBCT-vision treatment. The primary outcome is to compare the severity of the visual symptoms on a 0 to 10 scale between the two groups.

DETAILED DESCRIPTION:
Visual Snow Syndrome (VSS) is a neurological condition where affected people see flickering dots across their whole visual field, & may have other symptoms such as light sensitivity, after-images, trailing of images, & tinnitus. Functional Magnetic Resonance Imaging (fMRI) studies in VSS have shown brain network dysregulation involving the visual pathway. There is currently no evidence-based validated treatment for VSS, therefore the current standard of care is no treatment.

This research trial is to test the treatment of an intensive mindfulness programme, using the Mindfulness Based Cognitive Therapy customised for visual symptoms (MBCT-vision) programme, for people with Visual Snow Syndrome. MBCT-vision is a group learning programme, where people meet once weekly for 8 weeks. During these once weekly sessions, they learn mindfulness practices. The group discussions about the mindfulness practices introduces cognitive behavioural skills. Participants are given daily home practices between these weekly group learning sessions. We completed a study (ClinicalTrials.gov identifier NCT04184726) showing MBCT-vision was a feasible treatment for VSS.

This clinical trial is a 'randomized controlled trial'(RCT), where the effectiveness of a treatment is evaluated by comparison between two groups. We are recruiting people with VSS. Participants will be randomly allocated to one of two groups: one group receives MBCT-vision; while another group received standard care only for 5 months. The second group is called a waiting-list control group, whereby after 5 months, they will receive MBCT-vision treatment. The study will be conducted from single centre at a tertiary care hospital and the MBCT-vision is delivered online.

The key outcome of interest is severity of Visual Snow Syndrome on a 0-10 visual analogue scale. Other outcome measures will be collected to understand the effect of MBCT-vision, including quality of life and psychological wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* People with VSS according to the ICHD-3 criteria; previously diagnosed by a Neurologist, Ophthalmologist or Neuro-Ophthalmologist

Exclusion Criteria:

* Patients with co-morbid conditions affecting vision
* Patients with a current severe depressive or psychotic episode as determined by the psychologist
* Patients with severe difficulties in emotional regulation as determined by the psychologist
* Patients unable to provide informed consent for participation
* Patients with insufficient understanding of spoken English (due to need to participate in group discussions)
* Patients who have previously completed MBCT or similar mindfulness interventions
* Persons aged <16 or >80 years

An exploratory sub-study on the change in metabolomics will recruit healthy controls, inclusion criteria:

Healthy Control Inclusion Criteria

* Family or household member of a similar age (+/- 8years) to a participant with VSS recruited into the MBCT-vision VSS RCT study
* Person with no symptoms of VSS
* Person who self-declares as fit and well with no current medical conditions including anxiety or migraine

Healthy Control Exclusion Criteria

* Person unable to provide informed consent
* Person with other co-morbid medical or psychological conditions
* Person aged <16 or >80years

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Severity of visual symptoms of Visual Snow Syndrome on a 0-10 VAS | 5 months
  Severity of VSS visual symptoms

SECONDARY OUTCOMES:
Psychological wellbeing on the World Health Organisation (WHO) wellbeing index scores | 5 months
  WHO-5 wellbeing index
Psychological distress on the Clinical Outcomes in Routine Evaluation (CORE-10) scores | 5-months
  CORE-10 scores
Impact of Visual Snow Syndrome symptoms on daily life on 0-10 scale | 5-months
  VSS impact
Work and Social Adjustment Scale | 5-months
  impact of VSS on work and social function

CONTACTS AND LOCATIONS:
Overall Officials: Sui Wong, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No
anonymised numeric data to be shared upon reasonable request from qualified researcher after review by Eye Research Governance and data transfer agreement